CLINICAL TRIAL: NCT07255625
Title: Investigation of the Efficacy of Balance Training Program Applied With Stroboscopic Glasses in Female Volleyball Players With Chronic Ankle Instability
Brief Title: Effect of Stroboscopic Balance Training on Chronic Ankle Instability in Volleyball Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Berivan Beril Kılıç, Asistant professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Chronic Ankle Instability
Keywords: chronic ankle instability; stroboscopic glasses; balance training; volleyball athletes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroboscopic Glassess Group (Experimental): The athletes assigned to Group A underwent an eight-week balance training program using stroboscopic glasses, conducted twice a week under the supervision of a physiotherapist.
  Interventions: Device: Balance training with stroboscopic glasses
- Control Group (Active Comparator): The athletes assigned to Group B underwent an eight-week traditional balance training program, conducted twice a week under the supervision of a physiotherapist.
  Interventions: Other: Traditional Balance Training

INTERVENTIONS:
Device: Balance training with stroboscopic glasses — Participants in Group A completed a supervised, multi-modal balance training program while wearing Senaptec stroboscopic glasses (Beaverton, Oregon), set to a duty cycle of 100 ms transparent followed by 150 ms opaque. The glasses use liquid crystal lenses that alternate between clear and nearly opaque states when electrically activated and can operate in both binocular and monocular modes, with settings adjustable via a Bluetooth application. The program, targeting static and dynamic balance in individuals with chronic ankle instability, consisted of six progressively challenging exercises performed indoors, barefoot, in small groups, lasting approximately 20 minutes per session, twice weekly for eight weeks. Exercises were completed in two sets with 30-second rests between exercises and 2-minute rests between sets, and progression was adjusted based on participant performance.
  Arms: Stroboscopic Glassess Group
Other: Traditional Balance Training — The intervention consisted of a supervised, multi-modal balance training program targeting differentaspects of static and dynamic balance for participants with chronic ankle instability. The program included six progressively challenging exercises, administered under the supervision of a physiotherapist. Each session lasted approximately 20 minutes, and participants completed two sessions per week for eight weeks.
  The training was conducted indoors, barefoot, in small groups, with exercises performed in two sets, including 30-second rests between exercises and 2-minute rests between sets. Progression was implemented according to participants' performance throughout the program.
  Arms: Control Group

SUMMARY:
Effect of Stroboscopic Balance Training on Chronic Ankle Instability in Volleyball Players

DETAILED DESCRIPTION:
Ankle sprains are among the most common injuries in both athletes and the general population. A large-scale systematic review reported that ankle sprains account for approximately 80% of injuries occurring among athletes in most sports. Among volleyball players, ankle sprains are the most prevalent injury, constituting about 41% of all volleyball-related injuries. In athletes, performing certain technical or sport-specific tasks that require attention, such as running, sudden changes of direction, or landing, is associated with an increased risk of ankle sprain. Approximately 20% of acute ankle sprains progress to chronic conditions. Chronic ankle sprains lead to serious proprioceptive dysfunctions, including deficits in joint position sense and delayed peroneal muscle reaction time, resulting in significant ankle instability and balance impairment. Balance training in individuals with chronic ankle instability is concerned with improving postural control and has been recognized as an effective therapeutic approach for this population. Although there is evidence supporting the effectiveness of balance training in improving sensorimotor deficits in individuals with chronic ankle instability, including static and dynamic postural stability, muscle strength, and reinjury rates, reliance on visual information remains unchanged after conventional rehabilitation. The inability of visual input to utilize somatosensory feedback from the ankle joint has been identified as a factor contributing to recurrent ankle sprains in these individuals. Conventional interventions for chronic ankle instability do not address the need to correct altered somatosensory deficits following an ankle sprain. Therefore, a specific treatment option focusing on this neurophysiological dysfunction would be beneficial for these patients. Kim et al. reported the effect of stroboscopic vision in reactivating visual input in individuals with chronic ankle instability. Stroboscopic vision involves the use of special glasses in which the lenses alternate between transparent and opaque at intervals of 100 milliseconds, thereby reducing visual feedback. Balance training with stroboscopic glasses offers a different approach compared to conventional balance training. Stroboscopic balance training is a technique aimed at manipulating visual perception. In this method, the stroboscopic glasses intermittently block light, affecting the brain's processing of visual information. Consequently, the brain must process seen objects less continuously and less clearly. Stroboscopic glasses make rapid movements and changing situations more difficult to perceive, thereby challenging the balance system further. Conventional balance training, on the other hand, involves methods used to improve static and dynamic balance skills. This training approach aims to strengthen the balance mechanism through the use of specialized balance devices, exercises, and techniques. For example, balance boards, balance pads, trampolines, and various movement exercises are commonly used tools in conventional balance training. This method works on factors such as muscle strength, postural control, and coordination to improve static and dynamic balance control. The main difference between balance training with stroboscopic glasses and conventional balance training is the use of glasses that manipulate visual perception. These glasses challenge the brain's processing, thereby providing greater stimulation to the balance mechanism. In contrast, conventional balance training uses general exercises and tools to improve balance skills and does not focus on altering visual perception. Stroboscopic glasses have previously been used to improve sports performance in baseball players with positive results. They have also been incorporated into rehabilitation programs for individuals with chronic ankle instability, demonstrating beneficial outcomes. Although chronic ankle instability is a common problem among volleyball players, to our knowledge, no study has investigated a rehabilitation program using stroboscopic balance training in female volleyball players with chronic ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* Were professional female volleyball players.
* Had a history of at least two episodes of pain and swelling in the same ankle.
* Experienced at least one ankle sprain within the last six months.
* Exhibited persistent symptoms during functional activities and were free from symptoms related to any previous lower-extremity injuries.
* Reported a feeling of instability in the ankle joint.
* Had no other lower-extremity musculoskeletal injuries in the past six months.

Exclusion Criteria:

* Reported any vestibular or balance-related dysfunction.
* Had any systemic disease.
* Experienced an acute ankle sprain within the past six weeks.
* Had a history of fractures in the lower extremities.

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance Assessments | From enrollment to the end of treatment at 8 weeks
  Y Balance Test
Dynamic Balance Assessments | From enrollment to the end of treatment at 8 weeks
  Performanze Balance System

SECONDARY OUTCOMES:
Vertical Jump Test | From enrollment to the end of treatment at 8 weeks
Single Leg Hop Test | From enrollment to the end of treatment at 8 weeks
Active Joint Position Sense | From enrollment to the end of treatment at 8 weeks
Functional Assessments - Foot and Ankle Ability Measure-Sports Subscale (FAAM-Sport) | From enrollment to the end of treatment at 8 weeks
Functional Assessments - Cumberland Ankle Instability Tool | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Fatih, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Anaforoglu Kulunkoglu B, Celik D. Reliability and Validity of the Turkish Version of Foot and Ankle Ability Measure for Patients With Chronic Ankle Disability. J Foot Ankle Surg. 2019 Jan;58(1):38-41. doi: 10.1053/j.jfas.2018.07.007. Epub 2018 Nov 15. PMID 30448187
- [Result] Goble DJ. Proprioceptive acuity assessment via joint position matching: from basic science to general practice. Phys Ther. 2010 Aug;90(8):1176-84. doi: 10.2522/ptj.20090399. Epub 2010 Jun 3. PMID 20522675
- [Result] Carcia CR, Martin RL, Drouin JM. Validity of the Foot and Ankle Ability Measure in athletes with chronic ankle instability. J Athl Train. 2008 Apr-Jun;43(2):179-83. doi: 10.4085/1062-6050-43.2.179. PMID 18345343
- [Result] Haynes T, Bishop C, Antrobus M, Brazier J. The validity and reliability of the My Jump 2 app for measuring the reactive strength index and drop jump performance. J Sports Med Phys Fitness. 2019 Feb;59(2):253-258. doi: 10.23736/S0022-4707.18.08195-1. Epub 2018 Mar 27. PMID 29589412
- [Result] Shaffer SW, Teyhen DS, Lorenson CL, Warren RL, Koreerat CM, Straseske CA, Childs JD. Y-balance test: a reliability study involving multiple raters. Mil Med. 2013 Nov;178(11):1264-70. doi: 10.7205/MILMED-D-13-00222. PMID 24183777
- [Result] Powden CJ, Hoch JM, Jamali BE, Hoch MC. A 4-Week Multimodal Intervention for Individuals With Chronic Ankle Instability: Examination of Disease-Oriented and Patient-Oriented Outcomes. J Athl Train. 2019 Apr;54(4):384-396. doi: 10.4085/1062-6050-344-17. Epub 2018 Dec 27. PMID 30589387
- [Result] Gribble PA, Delahunt E, Bleakley CM, Caulfield B, Docherty CL, Fong DT, Fourchet F, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino W, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Athl Train. 2014 Jan-Feb;49(1):121-7. doi: 10.4085/1062-6050-49.1.14. Epub 2013 Dec 30. PMID 24377963
- [Result] Lee H, Han S, Hopkins JT. Altered Visual Reliance Induced by Stroboscopic Glasses during Postural Control. Int J Environ Res Public Health. 2022 Feb 12;19(4):2076. doi: 10.3390/ijerph19042076. PMID 35206263
- [Result] Kim KM, Estudillo-Martinez MD, Castellote-Caballero Y, Estepa-Gallego A, Cruz-Diaz D. Short-Term Effects of Balance Training with Stroboscopic Vision for Patients with Chronic Ankle Instability: A Single-Blinded Randomized Controlled Trial. Int J Environ Res Public Health. 2021 May 18;18(10):5364. doi: 10.3390/ijerph18105364. PMID 34069907
- [Result] Clark JF, Ellis JK, Bench J, Khoury J, Graman P. High-performance vision training improves batting statistics for University of Cincinnati baseball players. PLoS One. 2012;7(1):e29109. doi: 10.1371/journal.pone.0029109. Epub 2012 Jan 19. PMID 22276103
- [Result] Kim KM, Kim JS, Grooms DR. Stroboscopic Vision to Induce Sensory Reweighting During Postural Control. J Sport Rehabil. 2017 Sep 1;26(5). doi: 10.1123/jsr.2017-0035. Epub 2017 Jun 12. PMID 28605310
- [Result] Hertel J. Sensorimotor deficits with ankle sprains and chronic ankle instability. Clin Sports Med. 2008 Jul;27(3):353-70, vii. doi: 10.1016/j.csm.2008.03.006. PMID 18503872
- [Result] Song K, Rhodes E, Wikstrom EA. Balance Training Does Not Alter Reliance on Visual Information during Static Stance in Those with Chronic Ankle Instability: A Systematic Review with Meta-Analysis. Sports Med. 2018 Apr;48(4):893-905. doi: 10.1007/s40279-017-0850-8. PMID 29288435
- [Result] Song K, Burcal CJ, Hertel J, Wikstrom EA. Increased Visual Use in Chronic Ankle Instability: A Meta-analysis. Med Sci Sports Exerc. 2016 Oct;48(10):2046-56. doi: 10.1249/MSS.0000000000000992. PMID 27635773
- [Result] Molla-Casanova S, Ingles M, Serra-Ano P. Effects of balance training on functionality, ankle instability, and dynamic balance outcomes in people with chronic ankle instability: Systematic review and meta-analysis. Clin Rehabil. 2021 Dec;35(12):1694-1709. doi: 10.1177/02692155211022009. Epub 2021 May 31. PMID 34058832
- [Result] Hertel J. Functional instability following lateral ankle sprain. Sports Med. 2000 May;29(5):361-71. doi: 10.2165/00007256-200029050-00005. PMID 10840868
- [Result] Verhagen EA, Van der Beek AJ, Bouter LM, Bahr RM, Van Mechelen W. A one season prospective cohort study of volleyball injuries. Br J Sports Med. 2004 Aug;38(4):477-81. doi: 10.1136/bjsm.2003.005785. PMID 15273190
- [Result] Fong DT, Hong Y, Chan LK, Yung PS, Chan KM. A systematic review on ankle injury and ankle sprain in sports. Sports Med. 2007;37(1):73-94. doi: 10.2165/00007256-200737010-00006. PMID 17190537
- [Result] Chinn L, Hertel J. Rehabilitation of ankle and foot injuries in athletes. Clin Sports Med. 2010 Jan;29(1):157-67, table of contents. doi: 10.1016/j.csm.2009.09.006. PMID 19945591